CLINICAL TRIAL: NCT01996514
Title: Effect of Food Advertisements on Satiety and Meal-Time Food Intake in 9-14 y Old Boys and Girls
Brief Title: Food Advertisements, Satiety and Food Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FoodAdsKids_21595; MOP-82728 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Obesity Prevention
Keywords: Children; Food advertisement; Obesity; Television viewing; Food intake
MeSH Terms: conditions — Obesity | interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sweetener, non-food advertisements (Experimental): non-caloric sweetener with water followed by TV program with non-food advertisements while feeding at 30 min
  Interventions: Dietary Supplement: non-caloric sweetener with water; Behavioral: TV program with non-food advertisements while feeding
- Glucose, non-food advertisements (Experimental): Glucose with water followed by TV program with non-food advertisements while feeding at 30 min
  Interventions: Dietary Supplement: Glucose with water; Behavioral: TV program with non-food advertisements while feeding
- Sweetener, food advertisements (Experimental): non-caloric sweetener with water followed by TV program with food advertisements while feeding at 30 min
  Interventions: Dietary Supplement: non-caloric sweetener with water; Behavioral: TV program with food advertisements while feeding
- Glucose, food advertisements (Experimental): Glucose with water followed by TV program with food advertisements while feeding at 30 min
  Interventions: Dietary Supplement: Glucose with water; Behavioral: TV program with food advertisements while feeding

INTERVENTIONS:
Dietary Supplement: Glucose with water — Glucose (1.0 g•kg-1 body weight ) in 250 mL of water 30 min before meal
  Arms: Glucose, food advertisements; Glucose, non-food advertisements
Dietary Supplement: non-caloric sweetener with water — 0.15 g of the high-intensity sweetener, Splenda sucralose in 250 mL of water 30 min before meal
  Arms: Sweetener, food advertisements; Sweetener, non-food advertisements
Behavioral: TV program with non-food advertisements while feeding — 30 minutes of TV program containing non-food ads during a meal
  Arms: Glucose, non-food advertisements; Sweetener, non-food advertisements
Behavioral: TV program with food advertisements while feeding — 30 minutes of TV program containing non-food ads during a meal
  Arms: Glucose, food advertisements; Sweetener, food advertisements

SUMMARY:
We hypothesized that FA in a TV program watched during a meal, would block satiety responses to pre-meal energy consumption and delay satiation in OW/OB but not in NW boys and girls. Food intake was measured at 30 min following a glucose (1 g of glucose/kg body weight) or sweetened noncaloric beverage with or without the presence of food advertisements. Subjective appetite will be measured as well.

ELIGIBILITY:
Inclusion Criteria:

* born at full-term and of normal birth weight with no emotional, behavioral or learning problems

Exclusion Criteria:

* emotional, behavioral or learning problems dieting

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Food intake | at 30 min after treatment

SECONDARY OUTCOMES:
Subjective appetite | 0 to 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada